CLINICAL TRIAL: NCT03144947
Title: Phase II, Open Label, Randomized, Biomarker Study of Immune-mediated Mechanism of Action of Neoadjuvant Subcutaneous (SC) Trastuzumab in Patients With Operable or Locally Advanced/Inflammatory HER2-positive Breast Cancer (ImmunHER)
Brief Title: Biomarker Study of Immune-mediated Mechanism of Action of Neoadjuvant Trastuzumab in HER2+ Breast Cancer Patients
Acronym: IMMUN-HER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: University Hospital of Parma: Department of Biomedical, Biotechnological and Translational Sciences, Pathological Anatomy and Histology Unit (Unknown); University Hospital of Parma:Laboratory of Viral Immunopathology, Unit of Infectious Diseases and Hepatology (Unknown); University Hospital of Parma:Statistica medica ed epidemiologia clinica-UO Ricerca e Innovazione (Unknown); Clirest s.r.l. (Other); Mipharm SpA (Unknown); Arithmos srl (Unknown); Temas srl (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GOIRC-01-2016
Record Dates: First submitted 2017-04-07; First posted 2017-05-09 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cancer, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Non comparative, multi-center, open-label, neoadjuvant, randomized study, the purpose of randomization is to reduce bias owing to patient selection into treatments groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Trastuzumab IV (8 mg/kg loading dose, followed by 6 mg/kg) plus pertuzumab IV (840 mg loading dose, followed by 420 mg) plus docetaxel (75 mg/m2)*, every 3 weeks for 4 cycles.
  After surgery, study patients will receive trastuzumab IV x 14 cycles
  Interventions: Biological: Trastuzumab IV; Biological: Pertuzumab; Drug: Docetaxel
- Group B (Experimental): Trastuzumab SC (fixed dose of 600 mg) plus pertuzumab IV (840 mg loading dose, followed by 420 mg) plus docetaxel (75 mg/m2)*, every 3 weeks for 4 cycles. After surgery, study patients will receive trastuzumab SC x 14 cycles
  Interventions: Biological: Trastuzumab SC; Biological: Pertuzumab; Drug: Docetaxel

INTERVENTIONS:
Biological: Trastuzumab IV — Pre-randomization phase:
  FEC (fluorouracil 500 mg/m2; epirubicin 75 mg/m2; cyclophosphamide 500 mg/m2) x 3 cycles
  Post-randomization phase:
  Group A: Trastuzumab IV (8 mg/kg loading dose, followed by 6 mg/kg) plus pertuzumab IV (840 mg loading dose, followed by 420 mg) plus docetaxel (75 mg/m2)*, every 3 weeks for 4 cycles.
  by 420 mg) plus docetaxel (75 mg/m2)*, every 3 weeks for 4 cycles.
  *The dose of docetaxel may be escalated to 100 mg/m 2 at the investigator's discretion on subsequent cycles if the initial dose is well tolerated. After surgery, study patients will receive trastuzumab x 14 cycles using the same formulation (SC or IV) of the preoperative phase.
  Other Names: Herceptin-150 mg
  Arms: Group A
Biological: Trastuzumab SC — Pre-randomization phase:
  FEC (fluorouracil 500 mg/m2; epirubicin 75 mg/m2;
  Group B: Trastuzumab SC (fixed dose of 600 mg) plus pertuzumab IV (840 mg loading dose, followed by 420 mg) plus docetaxel (75 mg/m2)*, every 3 weeks for 4 cycles.
  *The dose of docetaxel may be escalated to 100 mg/m 2 at the investigator's discretion on subsequent cycles if the initial dose is well tolerated. After surgery, study patients will receive trastuzumab x 14 cycles using the same formulation (SC or IV) of the preoperative phase.
  Other Names: Herceptin-600 mg/5 mL
  Arms: Group B
Biological: Pertuzumab — pertuzumab IV (840 mg loading dose, followed by 420 mg) weeks for 4 cycles (both arms)
  Other Names: PerJeta 420 mg
Drug: Docetaxel — docetaxel (75 mg/m2), every 3 weeks for 4 cycles (both arms). The dose of docetaxel may be escalated to 100 mg/m2 at the investigator's discretion on subsequent cycles if the initial dose is well tolerated.
  Other Names: Docetaxel 20 MG/ML

SUMMARY:
Phase II, Open Label, Randomized, Biomarker Study of Immune-mediated Mechanism of Action of Neoadjuvant Subcutaneous (SC) Trastuzumab in Patients with Operable or Locally Advanced /Inflammatory HER2-positive Breast Cancer (ImmunHER)

DETAILED DESCRIPTION:
Women with histologically confirmed HER2-positive breast cancer with locally advanced, inflammatory,or early stage tumor (either greater than 2 cm in diameter or node positive) with no evidence of metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, infiltrating primary breast cancer with locally advanced, inflammatory, or early stage tumor (either greater than 2 cm in diameter or node positive) with no evidence of metastatic disease.
* HER2 positivity (either immunohistochemistry 3+ or fluorescent in situ hybridization amplification).
* Age 18 or older.
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* Availability of tumor tissue for biologic and molecular examination before starting primary treatment.
* Left ventricular ejection fraction within the institutional range of normal.
* Normal organ and marrow function.
* Adequate contraception methods for women of childbearing potential.
* Prior diagnosis of cancer is allowed as long as patient is free of disease and has been off treatment for the prior malignancy for a minimal interval of 3 years.
* Written informed consent.

Exclusion Criteria:

* Either stage I or IV breast cancer.
* Prior trastuzumab or pertuzumab.
* Any prior chemotherapy.
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment.
* Undergone major surgery (e.g., intrathoracic, intra-abdominal or intra-pelvic) 4 weeks prior to starting study drug or who have not recovered from side effects of such surgery.
* Breast radiotherapy prior to starting study.
* Known hypersensitivity to the investigational drugs or any of their excipients.
* Evidence of any disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an GOIRC-01-2016 ImmunHER Protocol Version 1.0, 11 April 2016 Page 6 of 140 investigational drug, or puts the patient at high risk for treatment-related complications.
* Moderate/severe hepatic impairment (Child- Pugh B/C).
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Concurrent malignancy or malignancy within 3 years prior to study enrollment, with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or insitu carcinoma of the uterine cervix.
* Pregnancy or breastfeeding (breast feeding should be discontinued to be enrolled in the study).
* Women of childbearing potential that refusal to adopt adequate contraceptive measures.
* Unwilling or unable to comply with the protocol. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2016-11-29 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Tumor Infiltrating lymphocites (TIL) rate on residual disease after either IV trastuzumab or SC trastuzumab (see related paragraph) | 6 months after last patient in
  stromal lymphocytes will be scored quantitatively on H&E stained whole-tumor slides as a continuous variable expressed as stromal percentage area within the tumor boundaries. For tumors with heterogeneous TILs, median values will be calculated from multiple counts from different tumor areas. Intra-epithelial TILs will also be recorded as well as tertiary lymphoid structures. Tumor regression will be scored based on recommended criteria.

SECONDARY OUTCOMES:
Associations between biomarkers (TIL, Tumor specific lymphocyte cell activity (TLA), and Fc-gamma-R polymorphisms) and between each biomarker with clinical outcome variables. | at baseline, 6 months and 5 years after last patient in
Frequency of toxicity Events: frequency of moderate and severe toxicity events and drop-out rate due to theraphy related toxicity (NCICommon Toxicity Criteria v 4.0) | 3.5 years
HRQOL during study treatment based on FACT-B | at baseline, and 6 months after last patient in
  mean FACT-B scores assessed at enrolment and mean FACT-B scores assessed before surgery.
Complete pathological response rate by treatment arm | 6 months after last patient in
5-year disease-free survival by treatment arm between treatment arms | 5 years

CONTACTS AND LOCATIONS:
Locations (21):
- Italy (21):
  - UO di Oncologia Ematologia, Azienda Ospedaliero Universitaria di Ferrara, Cona, Ferrara
  - UOC Oncologia Medica, Azienda ULSS21 di Legnago, Legnago, Verona
  - Oncologia Medica, Ospedale Sacro Cuore - Don Calabria - Negrar (VR), Negrar, Verona
  - UOC Oncologia-A.O. PAPA GIOVANNI XXIII Bergamo, Bergamo
  - SSD di Oncologia Medica Addarii, Policlinico S. Orsola-Malpighi,, Bologna
  - UOC di Oncologia. Azienda USL di Bologna, Ospedale Bellaria,, Bologna
  - Divisione di Oncologia Medica - Ospedale di Bolzano,, Bolzano
  - Breast Unit Spedali Civili di Brescia, Brescia
  - Investigational Clinical Oncology - INCOIRCCS-Fondazione del Piemonte per l'Oncologia (FPO), Candiolo
  - Chirurgia generale ad indirizzo senologico-Breast Unit Azienda Istituti Ospitalieri di Cremona, Cremona
  - Dipartimento di Medicina Interna e Specialità Mediche (DI.M.I.)-Università di Genova Clinica di Medicina Interna ad indirizzo oncologico, Genova
  - Oncologia Medica, IRST. Istituto Scientifico Romagnolo per lo studio e la cura dei Tumori, IRCCS di Meldola, Meldola (FC)
  - Dipartimento di Scienze Mediche e Chirurgiche, Materno Infantili e dell'adulto. Policlinico di Modena, Modena
  - SC di Oncologia Medica, A.O. San Gerardo, Monza
  - Azienda Ospedaliero-Universitaria di Parma, UOC di Oncologia Medica, Parma
  - Dipartimento di Oncologia e Ematologia, UO di Oncologia Medica Azienda USL di Piacenza, Piacenza
  - Struttura Complessa di OncologiaIRCCS- Istituto in Tecnologie Avanzate e Modelli Assistenziali in Oncologia Arcispedale Santa Maria Nuova, Reggio Emilia
  - UO di Oncologia. Azienda USL di Rimini, Rimini
  - Day Hospital, Ospedale di Sassuolo, Sassuolo
  - U.O. di Oncologia Medica PO "S. Chiara", Trento
  - Oncologia Medica Az. Ospedaliera di Verona, Verona

REFERENCES:
- [Derived] Pellegrino B, Tommasi C, Serra O, Gori S, Cretella E, Ambroggi M, Frassoldati A, Bisagni G, Casarini C, Bria E, Carbognin L, Fiorio E, Mura A, Zamagni C, Gianni L, Zambelli A, Montemurro F, Tognetto M, Todeschini R, Missale G, Campanini N, Silini EM, Maglietta G, Musolino A. Randomized, open-label, phase II, biomarker study of immune-mediated mechanism of action of neoadjuvant subcutaneous trastuzumab in patients with locally advanced, inflammatory, or early HER2-positive breast cancer-Immun-HER trial (GOIRC-01-2016). J Immunother Cancer. 2023 Nov 28;11(11):e007667. doi: 10.1136/jitc-2023-007667. PMID 38016718